CLINICAL TRIAL: NCT02870985
Title: BIOTRONIK-Safety and Clinical PerFormance of the Drug ELuting Orsiro Stent in the Treatment of Subjects With de Novo Coronary Artery Lesions-VI
Brief Title: BIOTRONIK Orsiro Pre-Marketing Registration
Acronym: BIOFLOW-VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik (Beijing) Medical Device Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C1207
Record Dates: First submitted 2016-08-05; First posted 2016-08-18 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIOTRONIK Orsiro SES (Experimental): Preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted. The procedure begins once percutaneous access has been made.Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed according to the QCA corelab guidelines.The subjects randomized to the experimental arm will be implanted with BIOTRONIK sirolimus eluting coronary stent(Orsiro).
  Interventions: Device: Coronary Stent
- Abbott Xience Prime™ EES (Active Comparator): Preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted. The procedure begins once percutaneous access has been made.Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed according to the QCA corelab guidelines.The subjects randomized to the comparator arm will be implanted with Abbott everolimus eluting coronary stent(Xience Prime™).
  Interventions: Device: Coronary Stent

INTERVENTIONS:
Device: Coronary Stent
  Other Names: percutaneous coronary intervention

SUMMARY:
The clinical investigation is a non-inferiority, multicenter, blinding evaluation, randomized, parallel controlled clinical study enrolling up to 440 subjects. All subjects will be randomized 1:1 to receive the BIOTRONIK Orsiro SES or the Abbott Xience Prime™ EES, in order to evaluate the efficacy and safety of the SES drug eluting stent in the treatment of coronary artery disease.

DETAILED DESCRIPTION:
Clinical or call follow up visits will take place at 1, 6, 12, 24, 36, 48 and 60 months post procedure. At 9 months (+ 30 days) all subjects will undergo a standard quantitative coronary angiography (QCA) follow up to assess the in-stent LLL as the main efficacious evaluation. Use the major adverse cardiac event (death, myocardial infarction and stent thrombosis) within one year post procedure as the main safety indicators to evaluate the investigational product's safety. The clinical and angiographic data sorting, calculation and statistical analysis will be conducted by an independent data management center and angiographic core laboratory.

ELIGIBILITY:
Inclusion Criteria-Clinical

1. Subject who can understand the investigation's goal has provided written informed consent, and is willing to comply with the study's follow-up requirements.
2. Subject is ≥ 18 years and ≤ 75 years old, male or female without pregnant.
3. Subject is an acceptable candidate for PCI.
4. Subject has clinical evidence of asymptomatic ischemia, stable or unstable angina pectoris or old myocardial infarction.
5. Subject has no contraindication for dual anti-platelet therapy treatment.

Inclusion Criteria-Angiographic

1. Target lesion must be in the major coronary artery or a branch (target vessel).
2. Target lesion must have angiographic evidence of ≥ 70% and < 100% stenosis (by operator's visual estimate).
3. Subject has up to two target lesions (two target lesions in one target vessel, or for each target vessel, it has one target lesion).
4. Target lesion is suitable for drug-eluting stent PCI treatment.
5. Target lesion must be ≤ 36 mm in length by operator's visual estimate, and can be completely covered by one stent.
6. Target vessel must have a reference vessel diameter of 2.25-4.0 mm by operator's visual estimate.
7. Target vessel must have a Thrombolysis In Myocardial Infarction (TIMI) flow ≥ 2.

Exclusion Criteria-Clinical

1. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
2. Subject has clinical symptoms and/or ECG changes consistent with acute ST elevation MI (STEMI) within 7 days prior to the index procedure, including hemodynamically unstable non-STEMI (NSTEMI) subjects.
3. Subject is hemodynamically unstable.
4. Subject is an unacceptable candidate for CABG.
5. Subject has a known allergy to contrast medium that cannot be adequately pre-medicated, or any known allergy to thienopyridine, aspirin, both heparin and bivalirudin, L-605 cobalt-chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten and nickel), acrylic, fluoropolymers, silicon carbide, PLLA, sirolimus or everolimus.
6. Previous revascularization of any target or non-target vessel 9 months prior to the index procedure.
7. Planned surgery within 6 months of the index procedure.
8. Planned staged treatment during the index procedure or within 30 days after the index procedure.
9. History of a stroke or transient ischemic attack (TIA) within 12 months prior to the index procedure.
10. Subjects with active bleeding disorders, active coagulopathy, or any other reason, who are ineligible for DAPT.
11. Subject will refuse blood transfusions.
12. Subject has documented severe cardiac failure (over III level of NYHA) or left ventricular ejection fraction (LVEF) ≤ 40% as evaluated by echocardiogram, left ventricular angiography, radionuclide ventriculography or any non-invasive imaging method within 90 days prior to the index procedure.
13. Subject is dialysis-dependent.
14. Subject has impaired renal function (i.e., creatinine > 2.0 mg/dL or 175 μmol/L determined) within 7 days prior to the index procedure.
15. Subject has leukopenia (i.e. WBC < 3.5*10*9/L), thrombocytopenia (plt<100*10*9/L) or thrombocytosis (PLT>350*10*9/L).
16. Subject is receiving chronic anticoagulation (e.g. coumadin, dabigatran, apixaban, rivaroxaban or any other agent).
17. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are excluded), or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; diabetes mellitus is excluded).
18. Subject has a life expectancy of < 3 years.
19. In the investigator's opinion, subject will not be able to comply with the follow-up requirements.
20. Subject is participating in another (medical device or drug) clinical study. Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.

Exclusion Criteria-Angiographic

1. Target lesion is located within a saphenous vein graft or arterial graft.
2. Target lesion has any of the following characteristics:

   1. Lesion location is within the left main coronary artery, or within 3 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX).
   2. Involves a side branch of > 2.5 mm in diameter. Note: Lesions within 3 mm of the origin of the right coronary artery may be treated.
3. Target lesion is totally occluded (100% stenosis).
4. Target vessel has angiographic evidence of thrombus.
5. Target vessel/lesion is excessively tortuous/angulated or is severely calcified, preventing complete inflation of an angioplasty balloon.
6. Target vessel was treated with brachytherapy at any time prior to the index procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Jing Xu, Principal Investigator — Tianjin Chest Hospital; Jian Zhang, Principal Investigator — TEDA International Cardiovascular Hospital; Yaling Han, Principal Investigator — General Hospital of Shenyang Military Region; Bo Yu, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Dan Song, Principal Investigator — Wuhan Asian Heart Hospital; Wen Xie, Principal Investigator — Teaching Hospital of Chengdu University of T.C.M.; Hui Li, Principal Investigator — Daqing oilfield general hospital; Ye Zhu, Principal Investigator — West China Hospital; Guosheng Fu, Principal Investigator — Sir Run Run Shaw Hospital; Biao Xu, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Urban P, Gershlick AH, Guagliumi G, Guyon P, Lotan C, Schofer J, Seth A, Sousa JE, Wijns W, Berge C, Deme M, Stoll HP; e-Cypher Investigators. Safety of coronary sirolimus-eluting stents in daily clinical practice: one-year follow-up of the e-Cypher registry. Circulation. 2006 Mar 21;113(11):1434-41. doi: 10.1161/CIRCULATIONAHA.104.532242. Epub 2006 Mar 13. PMID 16534015
- [Derived] Li C, Yang Y, Han Y, Song D, Xu J, Guan C, Gao R, Garcia-Garcia HM, Waksman R, Xu B; BIOFLOW VI Trial Investigators. Comparison of the Ultrathin Strut, Biodegradable Polymer Sirolimus-eluting Stent With a Durable Polymer Everolimus-eluting Stent in a Chinese Population: The Randomized BIOFLOW VI Trial. Clin Ther. 2020 Apr;42(4):649-660.e9. doi: 10.1016/j.clinthera.2020.02.014. Epub 2020 Apr 5. PMID 32268942
- See also: This link is a PubMed URL that allows you to view an article about the efficacy and safety of high-frequency stimulation in patients with atrial fibrillation: a randomized controlled trial. PubMed is a free resource that supports the search and retrieval — http://www.ncbi.nlm.nih.gov/pubmed?term=16534015%5Buid%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: July 2015 - September 2016 totally 11 investigational sites(hospitals) in China
Period: Overall Study
Arm/Group | Abbott Xience Prime™ EES | BIOTRONIK Orsiro SES
Started | 220 | 220
Completed | 220 | 220
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The subjects have been randomized and implanted with Abbott Xience Prime™ EES or BIOTRONIK Orsiro SES
Groups:
- Total: Total of all reporting groups
Arm/Group | Abbott Xience Prime™ EES | BIOTRONIK Orsiro SES | Total
Number analyzed (Participants) | 220 | 220 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.38 (8.62) | 59.05 (8.48) | 58.715 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 60 | 138
  Male | 142 | 160 | 302
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 220 | 220 | 440

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Lumen Loss at 9 Months as Assessed by the Core Laboratory QCA Analysis
Description: QCA data will be provided by an independent core laboratory. A separate report with descriptive statistics will be provided by the core laboratory in accordance with their guidelines.
  For the primary endpoint, both the lesion and patient level analysis will be done for 9-month in-stent LLL. The analysis on patient level for FAS is considered as main analysis. Other analysis based on lesion level and/or PPS is only for supportive purposes.
Time Frame: At 9 months post procedure
Population: There were 220 subjects who conducted the procedure in each group.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- BIOTRONIK Orsiro SES: Patients implanted with Orsiro SES stents of BIOTRONIK
- Abbott Xience Prime™ EES: Patients implanted with Xience Prime™ EES stents of Abbot Laboratories
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 220 | 220
mm | 0.05 (0.21) | 0.07 (0.22)

2. Secondary Outcome: Number of Participants With Main Adverse Cardiac Event (MACE)
Description: Main adverse cardiac event include all-cause death, Q wave or non-Q wave myocardial infarction and clinically driven TLR.
  The comparison between the two treatment groups for the secondary endpoints will be presented by the same anaysis method as baseline characteristics.
  The normally distributed quantitative variables will be compared by Student's t-test and the qualititative vairiables which are not normally distributed will be compared by using Wilcoxon sum-rank test.
Time Frame: At 5 years post-procedure
Population: There were 216 subjects who conducted the procedure and finished the 5 years following up in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 216 | 216
Participants | 17 | 13

3. Secondary Outcome: Number of Participants With All-cause Death
Description: The MACEs in the test group included 6 cases of all-cause death.Among them:
  1. One subject died from upper gastrointestinal hemorrhage, which had no obvious relation to the operation and device.
  2. Two subjects died from gastric cancer and COVID-19 complicated with respiratory failure respectively, which was unrelated to the operation and device.
  3. One subject died suddenly at home on Day 192 after the baseline operation, with the cause of death unknown.
  4. During the 3-year follow-up, subject family member told that he/she had ever been hospitalized for cardiac failure, but died after invalid rescue. The event was determined as cardiac death, of which the relationship with the operation and device cannot be determined.
  5. During the 3-year follow-up of another subject, his/her family member told that he/she had died. For which his/her family member was reluctant to provide relevant supporting documents, the relationship with the operation and device cannot be determined.
Time Frame: At 5 years post-procedure
Population: There were 216 subjects who conducted the procedure and finished the 5 years following up in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 216 | 216
Participants | 6 | 6

4. Secondary Outcome: Number of Participants With Cardiac Death
Description: Two subjects with Cardica death in test group:
  1. One of the patient died of sudden death at home, with the cause of death unknown.The patient participated in the trial on April 15, 2016. He/She was treated in local hospital for chest tightness and syncope in September 2016. He was considered to have rheumatic heart disease, heart failure and cardiogenic syncope. After treatment, he was improved and discharged from hospital and died in October 2016. The possibility of sudden cardiac death caused by ventricular arrhythmia cannot be excluded.
  2. During the 3-year follow-up of a subject, his/her family member told that he/she had ever been hospitalized for cardiac failure, but the subject eventually died after invalid rescue of cardiac failure. As the hospital did not have definite basis for acute myocardial infarction during the event. Therefore, the event was determined as cardiac death, of which the relationship with the operation and device cannot be determined.
Time Frame: At 5 years post-procedure
Population: There were 216 subjects who conducted the procedure and finished the 5 years following up in each group.
Measure: Count of Participants; unit: Participants
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 216 | 216
Participants | 2 | 0

5. Secondary Outcome: Number of Participants With Myocardial Infarction
Description: Including Q-wave and Non Q-wave myocardial infarction. The comparison between the two treatment groups for the secondary endpoints will be presented by the same anaysis method as baseline characteristics.
  The normally distributed quantitative variables will be compared by Student's t-test and the qualititative vairiables which are not normally distributed will be compared by using Wilcoxon sum-rank test.
Time Frame: At 5 years post-procedure
Population: 220 patients were enrolled in the each group. 5 patients died in the test group, and there was no myocardial infarction during the 5-year follow-up, and 4 patients were lost 5 follow-up. excluding these patients, the analysis population of the test group was 211.
  6 patients died in the test group, and there was no myocardial infarction during the 5-year follow-up, and 4 patients were lost 5 follow-up. excluding these patients, the analysis population of the test group was 210.
Measure: Count of Participants; unit: Participants
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 211 | 210
Participants | 7 | 3

6. Secondary Outcome: Number of Participants With TVR Myocardial Infarction
Description: Target vessel-related myocardial infarction
Time Frame: At 5 years post-procedure
Population: 4 subjects lost contact in each group at 5 years of follow-up. In the test group, 5 subjects dead, and no happened TVR myocardial infarction, Except for these subjects, the analysis population of the test group is 211.
  In the control group, 6 subjects dead, and no happened TVR myocardial infarction. Except for these subjects, the analysis population of the control group is 210.
Measure: Count of Participants; unit: Participants
Groups:
- Abbott Xience Prime™ EES: Active Comparator: Abbott Xience Prime™ EES Preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted. The procedure begins once percutaneous access has been made.Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed according to the QCA corelab guidelines.The subjects randomized to the comparator arm will be implanted with Abbott everolimus eluting coronary stent(Xience Prime™).
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 211 | 210
Participants | 4 | 2

7. Secondary Outcome: In-stent Thrombus
Description: During the 5-year clinical follow-up after baseline operation, one stent thrombosis event occurred in the test group. On July 21, 2016, the subject was implanted with the Orsiro Sirolimus-Eluting Coronary Stent System due to coronary heart disease. As the subject developed chest pain again, the coronary angiography reexamination was performed on March 22, 2019. During the operation, the OCT (optical coherence tomography) showed stent thrombosis in the right coronary artery, and then thrombus aspiration was performed. Investigators in the clinical trial center where the subject was enrolled believed that the stent thrombosis identified 972 days after the baseline operation belonged to very late stent thrombosis (VLST). The causes of its occurrence were considered to be related to the stent malapposition caused by insufficient stent expansion during the baseline operation and the possible platelet resistance of the subject.
Time Frame: At 5 years post-procedure
Population: 4 subjects lost contact in each group at 5 years of follow-up. In the test group, 5 subjects dead, and no happened In-stent thrombus, Except for these subjects, the analysis population of the test group is 211.
  In the control group, 6 subjects dead, and no happened In-stent thrombus. Except for these subjects, the analysis population of the control group is 210.
Measure: Count of Participants; unit: Participants
Groups:
- BIOTRONIK Orsiro SES: Experimental: BIOTRONIK Orsiro SES Preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted. The procedure begins once percutaneous access has been made.Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed according to the QCA corelab guidelines.The subjects randomized to the experimental arm will be implanted with BIOTRONIK sirolimus eluting coronary stent(Orsiro).
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 211 | 210
Participants | 1 | 0

8. Secondary Outcome: Number of Participants With TLR
Description: Target lesion revascularization
Time Frame: At 5 years post-procedure
Population: 4 subjects lost contact in each group at 5 years of follow-up. In the test group, 5 subjects dead, and no happened TLR, Except for these subjects, the analysis population of the test group is 211.
  In the control group, 6 subjects dead, and no happened TLR. Except for these subjects, the analysis population of the control group is 210.
Measure: Count of Participants; unit: Participants
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
Number analyzed (Participants) | 211 | 210
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: At 5 years post-procedure
Groups:
- BIOTRONIK Orsiro SES: Preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted. The procedure begins once percutaneous access has been made.Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed according to the QCA corelab guidelines.The subjects randomized to the experimental arm will be implanted with BIOTRONIK sirolimus eluting coronary stent(Orsiro).
  Coronary Stent
- Abbott Xience Prime™ EES: Preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted. The procedure begins once percutaneous access has been made.Following intracoronary injection of nitroglycerin or isosorbide dinitrate, a baseline angiography of the target vessel must be performed according to the QCA corelab guidelines.The subjects randomized to the comparator arm will be implanted with Abbott everolimus eluting coronary stent(Xience Prime™).
  Coronary Stent
Arm/Group | BIOTRONIK Orsiro SES | Abbott Xience Prime™ EES
All-Cause Mortality (participants affected / at risk) | 6/216 | 6/216
Serious Adverse Events (participants affected / at risk) | 82/216 | 79/216
Other Adverse Events (participants affected / at risk) | 148/216 | 141/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Orsiro SES (N=216) | Abbott Xience Prime™ EES (N=216)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 2 (2)
Type 2 diabetic patient (Gastrointestinal disorders) | 2 (2) | 2 (2)
Coronary heart disease (Cardiac disorders) | 10 (11) | 10 (10)
Cerebral infarction (Vascular disorders) | 6 (6) | 4 (4)
Gastric diseases (Gastrointestinal disorders) | 8 (9) | 7 (10) — Including gastric carcinoma, gastrorrhagia, gastroesophageal reflux, gastric ulcer, gastritis, gastrointestinal bleeding, etc...
Target lesion revascularization (Cardiac disorders) | 3 (4) | 4 (4)
Target vessel revascularization (Cardiac disorders) | 9 (10) | 13 (13)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Non-target vessel revascularization (Cardiac disorders) | 9 (9) | 8 (8)
Unstable angina pectoris (Cardiac disorders) | 11 (12) | 15 (22)
MI(myocardial infarction) (Cardiac disorders) | 6 (6) | 3 (3)
Post- PCI (Cardiac disorders) | 3 (4) | 9 (9)
Bosom frowsty chest pain (General disorders) | 3 (3) | 9 (10)
Heart related diseases (Cardiac disorders) | 11 (12) | 6 (6) — Including: Acute non-ST elevation myocardial infarction Exertional angina Old myocardial infarction arrhythmology Angina pectoris Heart failure Cardiac death Precardiac discomfort Cardiac insufficiency Atrial flutter Atrial tachycardia
Kidney related diseases (Renal and urinary disorders) | 7 (7) | 3 (4)
Other diseases (General disorders) | 24 (33) | 23 (26)
Dental related diseases (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (5) — Including: Bleeding gums Gingival bleeding epistaxis periodontitis Tooth mobility Periapical periodontitis Periodontal abscess
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Orsiro SES (N=216) | Abbott Xience Prime™ EES (N=216)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (4)
Type 2 diabetic patient (Gastrointestinal disorders) | 0 (0) | 4 (4)
Coronary heart disease (Cardiac disorders) | 8 (8) | 7 (7)
Cerebral infarction (Vascular disorders) | 2 (2) | 2 (2)
Gastric diseases (Gastrointestinal disorders) | 7 (9) | 4 (4) — Including: gastritis Gastric ulcer Chronic gastritis The gastric mucosa is congested Upset stomach Chronic non-atrophic gastritis with erosion Acute gastroenteritis
Chest tightness of chest pain (General disorders) | 54 (73) | 50 (63)
Troponin is elevated (Cardiac disorders) | 13 (14) | 18 (18)
hypohepatia (Hepatobiliary disorders) | 6 (6) | 3 (3)
Post-PCI (Cardiac disorders) | 12 (12) | 5 (5)
Have a headache giddy (General disorders) | 5 (5) | 3 (3)
unstable angina pectoris (Cardiac disorders) | 3 (3) | 7 (7)
Hypertension (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Heart related diseases (Cardiac disorders) | 13 (14) | 8 (8) — Including: The cause of palpitations is unknown Atrial tachycardia Stable angina pectoris tachycardia Sinus bradycardia Exertional angina Cardiac insufficiency arrhythmology
Kidney related diseases (Renal and urinary disorders) | 6 (6) | 6 (6) — Including: Blood in the urine hyperuricemia The cause of the painful urine is unknown Urinary tract infection The left kidney cyst Renal insufficiency Ureteral calculi prostatitis Left renal cyst prostatic hyperplasia
Other diseases (General disorders) | 47 (72) | 47 (67) — Mainly Including: High blood pressure esophagitis Room sex premature beat Lower blood pressure Allergic dermatitis Left knee joint trauma tenosynovitis upper respiratory tract infection (URTI) Gastrointestinal bleeding Subcutaneous bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02870985/Prot_SAP_000.pdf